CLINICAL TRIAL: NCT04408547
Title: Technical Factors of Embryo Transfer Procedure That Might Affect the Outcome
Acronym: IAFACT
Status: Completed | Type: Observational
Sponsor: Iakentro Fertility Centre (Other)
Responsible Party: Principal Investigator, Yannis Prapas, Professor of Obstetrics - Gynaecology, Iakentro Fertility Centre
Other Study IDs: IakentroFC
Record Dates: First submitted 2020-05-13; First posted 2020-05-29 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: IVF; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- soft catheter: Patients who underwent embryo transfer with a soft catheter
  Interventions: Device: embryo transfer catheter
- stiff catheter: Patients who underwent embryo transfer with a stiff catheter because soft couldn't pass
  Interventions: Device: embryo transfer catheter

INTERVENTIONS:
Device: embryo transfer catheter — undergoing embryo transfer

SUMMARY:
Analysis our Embryo transfer data, prospectively collected during the last 6 years (2014- 2019), performed by the same operator YP, who has been doing embryo transfers since 1984. All factors that might impact the embryo transfer will be analyzed. We want to see which factors that influence the success rate are not related to the subjectivity of the operator and could be adjusted through different approaches.

DETAILED DESCRIPTION:
Most patients undergoing IVF or ICSI reach a blastocyst embryo transfer but less achieve pregnancy and live birth. Many reasons have been proposed to explain these results. Among them, the factor Embryo Transfer Procedure gained less of the attention since few papers have been published and most of them had a lot of biases. In order to eliminate possible biases, we wanted to analyze our Embryo transfer data, prospectively collected during the last 6 years (2014- 2019), performed by the same operator YP, who has been doing embryo transfers since 1984. All factors that might impact the embryo transfer will be analyzed. We want to see which factors that influence the success rate are not related to the subjectivity of the operator and could be adjusted through different approaches.

Primary outcomes: bhCG positive rate, pregnancy rate, ongoing pregnancy rate, live birth rate.

Secondary outcomes: Full bladder, uterine ax orientation, Endometrial thickness, type of catheter, straightforward advancement of the preloaded catheter, use of a stiffer hard catheter to pass through the cervix and the orifice, the site of the uterine cavity that the embryo was released, single or double transfer due to blocked embryo in the catheter.

In addition for each embryo transfer variables that may influence the pregnancy rates will be collected: age of the woman, number of oocytes harvested, sperm characteristics, fertilization rate, stage and grade of the embryos the day of transfer

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing embryo transfer after IVF

Exclusion Criteria:

* Women with known embryo implantation issues

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women can undergo embryo transfer
Study Population: Women undergoing embryo transfer after IVF
Sampling Method: Non-Probability Sample
Enrollment: 3512 (Actual)
Dates: Start 2014-01-03 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with bhCG positive test after embryo transfer | Number of patients bhCG positive up to12 days after embryo transfer
  Number of patients bhCG positive up to12 days after embryo transfer
Number of patients with on going clinical pregnancy | Number of patients with on going clinical pregnancy up to 12 weeks after embryo transfer
  Number of patients with on going clinical pregnancy up to12 weeks after embryo transfer
Number of live births after embryo transfer | Number oflive birth up to 9 months after embryo transfer
  Number oflive birth up to9 months after embryo transfer

SECONDARY OUTCOMES:
Percentage of fullnes of bladder | At the time of embryo transfer and the impact of pregnancy test result 12 days after the mebryo transfer
  Percentage of fullness of the bladder during embryo transfer
Endometrial thickness | prior to embryo transfer
  Endometrial thickness prior to embryo transfer
Uterine axe orientation | At the time of embryo transfer and the impact of pregnancy test result 12 days after the mebryo transfer
  Uterine axe orientation during embryo transfer
Type of embryo transfer catheter | At the time of embryo transfer and the impact of pregnancy test result 12 days after the mebryo transfer
  Type of embryo transfer catheter used in the procedure
Distance from the fundus of the embryo release | At the time of embryo transfer and the impact of pregnancy test result 12 days after the mebryo transfer
  Distance from the fundus of the embryo release
Embryo retained in the catheter | Number of patients who underwent embryo transfer and the embryo was retained in the catheter at the time of embryo transfer and the impact of pregnancy test result 12 days after the mebryo transfer
  Embryo retained in the catheter

CONTACTS AND LOCATIONS:
Locations (1):
- IAKENTRO Fertility Center, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Prapas N, Prapas Y, Panagiotidis Y, Prapa S, Vanderzwalmen P, Makedos G. Cervical dilatation has a positive impact on the outcome of IVF in randomly assigned cases having two previous difficult embryo transfers. Hum Reprod. 2004 Aug;19(8):1791-5. doi: 10.1093/humrep/deh320. Epub 2004 Jun 3. PMID 15178658